CLINICAL TRIAL: NCT04499248
Title: A Phase 1/2 Study to Evaluate the Safety and Efficacy of AGN-193408 SR in Participants With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: AGN-193408 SR in the Treatment of Open-angle Glaucoma or Ocular Hypertension
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1833-201-407
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: Open-angle glaucoma; Ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1 -Dose A (Experimental): Single dose of AGN-193408 SR Dose A administered in the study eye on Day 1. One drop of Lumigan 0.01% administered in the non-study eye once daily every evening starting on Day 1.
  Interventions: Drug: AGN-193408 SR; Other: Lumigan
- Cohort 1 - Dose B (Experimental): Single dose of AGN-193408 SR Dose B administered in the study eye on Day 1. One drop of Lumigan 0.01% administered in the non-study eye once daily every evening starting on Day 1.
  Interventions: Drug: AGN-193408 SR; Other: Lumigan
- Cohort 2 - Dose A (Experimental): AGN-193408 SR Dose A (single dose on Day 1) + vehicle eye drops (once daily in the evening starting on Day 1) administered in the study eye. Lumigan (once daily in the evening starting on Day 1) + Sham AGN-193408 SR (single administration on Day 1) administered in the non-study eye.
  Interventions: Drug: AGN-193408 SR; Other: Lumigan; Other: Sham Administration; Other: Lumigan Vehicle
- Cohort 2 - Dose B (Experimental): AGN-193408 SR Dose B (single dose on Day 1) + vehicle eye drops (once daily in the evening starting on Day 1) administered in the study eye. Lumigan (once daily in the evening starting on Day 1) + Sham AGN-193408 SR (single administration on Day 1) administered in the non-study eye.
  Interventions: Drug: AGN-193408 SR; Other: Lumigan; Other: Sham Administration; Other: Lumigan Vehicle
- Cohort 3 - Dose A (Experimental): AGN-193408 SR Dose A (single dose on Day 1) + vehicle eye drops (once daily in the evening starting on Day 1) administered in the study eye. Lumigan (once daily in the evening starting on Day 1) + Sham AGN-193408 SR (single administration on Day 1) administered in the non-study eye.
  Interventions: Other: Lumigan; Drug: AGN-193408 SR; Other: Sham Administration; Other: Lumigan Vehicle
- Cohort 3 - Dose B (Experimental): AGN-193408 SR Dose B (single dose on Day 1) + vehicle eye drops (once daily in the evening starting on Day 1) administered in the study eye. Lumigan (once daily in the evening starting on Day 1) + Sham AGN-193408 SR (single administration on Day 1) administered in the non-study eye.
  Interventions: Other: Lumigan; Drug: AGN-193408 SR; Other: Sham Administration; Other: Lumigan Vehicle

INTERVENTIONS:
Drug: AGN-193408 SR — An implant containing preservative-free AGN-193408 dispersed in a biodegradable polymer matrix. Implants are preloaded into an applicator to facilitate insertion of the implant into the anterior chamber of the study eye.
  Arms: Cohort 1 - Dose B; Cohort 1 -Dose A; Cohort 2 - Dose A; Cohort 2 - Dose B
Other: Lumigan — Control Treatment in Fellow Eye Lumigan 0.01% is a topical eye drop that is a solution containing 0.1 mg/mL bimatoprost
  Other Names: Active Comparator
Other: Sham Administration — Needleless applicator contacting similar intracameral insertion location on eye as AGN-193408 SR.
  Arms: Cohort 2 - Dose A; Cohort 2 - Dose B
Other: Lumigan Vehicle — Vehicle eye drops (for masking) will be administered once daily in the evening starting on Day 1 in the study eye during Cohort 2.
  Other Names: Vehicle
  Arms: Cohort 2 - Dose A; Cohort 2 - Dose B
Drug: AGN-193408 SR — An implant containing preservative-free AGN-193408 dispersed in a biodegradable polymer matrix. Implants are preloaded into an applicator to facilitate insertion of the implant in the study eye.
  Arms: Cohort 3 - Dose A; Cohort 3 - Dose B
Other: Sham Administration — Needleless applicator contacting similar insertion location on eye as AGN-193408 SR.
  Arms: Cohort 3 - Dose A; Cohort 3 - Dose B
Other: Lumigan Vehicle — Vehicle eye drops (for masking) will be administered once daily in the evening starting on Day 1 in the study eye during Cohort 3.
  Other Names: Vehicle
  Arms: Cohort 3 - Dose A; Cohort 3 - Dose B

SUMMARY:
This is a multicenter, open-label, dose escalation (Cohort 1) to masked, randomized, parallel-groups (Cohort 2) and (Cohort 3) study to evaluate the safety and efficacy of AGN-193408 SR in participants with open-angle glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing to withhold his/her IOP (Intraocular Pressure) treatments according to the study requirements, and in the opinion of the investigator, can do so without significant risk.
* Diagnosis of either OAG [open-angle glaucoma] (ie, [POAG], pseudoexfoliation glaucoma,pigmentary glaucoma) or OHT (ocular hypertension) in both eyes.
* Must be pseudophakic (at least 4 months postcataract surgery prior to treatment administration [Cycle 1 Day 1 Administration visit]) (Cohort 3 only).

Exclusion Criteria:

* Known allergy or sensitivity to any study medication or its components, any component of the delivery vehicle, procedure-related materials, or diagnostic agents used during the study (eg, topical anesthetic, dilating drops, fluorescein, povidone-iodine).
* Concurrent or anticipated enrollment in an investigational drug or device study or participation in such a study within 2 months prior to the Baseline visit through the final study visit.
* History of intracameral implant in the study eye (eg, Bimatoprost SR, OTX-TIC, ENV515 Travoprost XR).
* History of laser trabeculoplasty within 6 months prior to screening in the study eye.
* History or evidence of clinically relevant, substantial ocular trauma (eg, a traumatic cataract, traumatic angle recession, etc.) in the study eye.
* History or evidence of complicated cataract/lens surgery, as stated in the protocol.
* Intraocular surgery (including cataract surgery) in the study eye within the 4 months prior to treatment administration.
* Any history of corneal graft, including partial grafts (eg, Descemet's Stripping Endothelial Keratoplasty [DSEK], Descemet's Membrane Endothelial Keratoplasty [DMEK]); or incisional refractive surgery (eg, radial keratotomy), other than astigmatic keratotomy or limbal relaxing incisions in the study eye.
* History of herpetic ocular diseases in either eye (including herpes simplex virus and varicella zoster virus).
* Anticipated need for any incisional or laser ocular surgery in either eye during the study.
* History of anatomically narrow angle resulting in evidence of angle changes or any history or closed angle glaucoma in the study eye.
* History or evidence of a peripheral iridotomy/iridectomy in the inferior iris in the study eye.
* Any history of trabeculectomy or other types of incisional glaucoma surgery, including a glaucoma seton or aqueous bypass stents in either eye, or minimally invasive glaucoma surgery (MIGS) type trabecular meshwork surgeries in the study eye.
* Anticipated use of corticosteroids in either eye except for permitted interventions or systemically during the study, or historical use prior to Baseline within:

  * 3 years: intraocular fluocinolone acetonide
  * 6 months: intraocular corticosteroid(s) other than fluocinolone; any injectable periocular or sub-Tenon's/subconjunctival corticosteroid
  * 2 months: systemic (eg, oral, intramuscular, intravenous) or topical ocular corticosteroids
  * 2 weeks: dermal corticosteroids applied to skin of the eyelid(s), around the eye, or adnexa.
* Anticipated use of other topical ocular medications in either eye except for permitted interventions.
* The anticipated wearing of contact lenses in the study eye (Cohort 1) and both eyes (Cohorts 2 and 3) during the study that deviates from the following (contact lens wear is allowed during the study, but is to be temporarily discontinued before study visits, and before and after an Administration Day according to the following):

  * Use of soft lenses should be discontinued at least 3 days prior to Baseline, and use of rigid gas permeable or hard contact lenses should be discontinued at least 1 week prior to Baseline
  * Use of soft lenses should be discontinued at least 3 days and use of rigid gas permeable or hard contact lenses should be discontinued at least 1 week prior to a scheduled study visit or Administration Day visit
  * Use of contact lenses of any kind should be discontinued for 1 week following any AGN-193408 SR administration
* Central corneal thickness of < 480 or > 620 micrometers in both eyes.
* Visual field loss in the study eye that, in the opinion of the investigator, is functionally significant (eg, split fixation, field defect within the central 10 degrees that is visually significant or likely to cause central visual impairment upon progression) or shows evidence of progressive visual field loss within the year prior to Baseline.
* Evidence of macular edema in either eye during screening or in participant's medical history.
* At Screening, evidence of posterior synechia behind the iris inferiorly in the study eye that in the investigator's opinion may inhibit the ability to safely receive at least 1 AGN-193408 SR implant (Cohort 3 only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hour 0 Intraocular Pressure (IOP) in the Study Eye | Baseline to Month 36
  IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Number of participants experiencing treatment emergent adverse events | Baseline to Month 36

SECONDARY OUTCOMES:
Time to Rescue Treatment or Re-Treatment in the Study Eye | Baseline to Month 36
  Time to rescue treatment or the second treatment is defined as the time between the first treatment and the second treatment in the study eye.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (49):
- United States (42):
  - Horizon Eye Specialists & Lasik Center - Sun City /ID# 252153, Sun City, Arizona
  - Global Research Management /ID# 241699, Glendale, California
  - United Medical Research Institute /ID# 241701, Inglewood, California
  - Lakeside Vision Center /ID# 241698, Irvine, California
  - The Eye Research Foundation /ID# 234528, Newport Beach, California
  - Sacramento Eye Consultants /ID# 241697, Sacramento, California
  - Premiere Practice Management LLC /ID# 235957, Torrance, California
  - Wolstan & Goldberg Eye Associates /ID# 241700, Torrance, California
  - Connecticut Eye Consultants P.C. /ID# 235862, Danbury, Connecticut
  - Brandon Eye Associates - Brandon /ID# 276600, Brandon, Florida
  - Nature Coast Clinical Research - Crystal River /ID# 237781, Crystal River, Florida
  - Advanced Research, LLC /ID# 276987, Deerfield Beach, Florida
  - University of Florida Health Ophthalmology - Jacksonville /ID# 243122, Jacksonville, Florida
  - East Florida Eye Institute /ID# 235762, Stuart, Florida
  - Logan Ophthalmic Research Inc. /ID# 252087, Tamarac, Florida
  - Coastal Research Associates /ID# 234649, Roswell, Georgia
  - Thomas Eye Group PC /ID# 266775, Sandy Springs, Georgia
  - University of Illinois Hospital and Health Sciences System /ID# 253630, Chicago, Illinois
  - Midwest Medical Advisors Inc /ID# 235845, Carmel, Indiana
  - Indiana University - Glick Eye Institute /ID# 235887, Indianapolis, Indiana
  - Ophthalmic Consultants of Boston /ID# 236535, Boston, Massachusetts
  - Fraser Eye Care Center /ID# 267100, Fraser, Michigan
  - Midwest Vision Research Foundation at Pepose Vision Institute /ID# 267094, Chesterfield, Missouri
  - Silverstein Eye Centers /ID# 266767, Kansas City, Missouri
  - Tekwani Vision Center /ID# 235149, St Louis, Missouri
  - Nv Eye Surgery - Henderson /ID# 276925, Henderson, Nevada
  - Rutgers New Jersey Medical School Campus, Doctors Office Center /ID# 234365, Newark, New Jersey
  - Northern New Jersey Eye Institute /ID# 241545, South Orange, New Jersey
  - Asheville Eye Associates /ID# 234963, Asheville, North Carolina
  - Private Practice - Dr. James D. Branch /ID# 234560, Winston-Salem, North Carolina
  - The Ohio State University /ID# 267590, Columbus, Ohio
  - Oklahoma Eye Surgeons /ID# 252089, Oklahoma City, Oklahoma
  - Drs Fine Hoffman & Sims LLC /ID# 235919, Eugene, Oregon
  - Scott and Christie and Associates /ID# 252284, Cranberry Township, Pennsylvania
  - Eye Specialty Group /ID# 252201, Memphis, Tennessee
  - Vanderbilt Eye Institute /ID# 266915, Nashville, Tennessee
  - Advancing Vision Research /ID# 236683, Smyrna, Tennessee
  - Macro Trials (SMO/Network/Consortium) /ID# 266772, Austin, Texas
  - San Antonio Eye Center /ID# 272087, San Antonio, Texas
  - St. George Eye Center /ID# 236200, St. George, Utah
  - Piedmont Eye Center /ID# 246455, Lynchburg, Virginia
  - Vistar Eye Center /ID# 234811, Roanoke, Virginia
- Japan (7):
  - Kitasato University Hospital /ID# 238880, Sagamihara-shi, Kanagawa
  - National Hospital Organization Saitama Hospital /ID# 266953, Wako, Saitama
  - Duplicate_Shimane University Hospital /ID# 238641, Izumo-shi, Shimane
  - The University of Tokyo Hospital /ID# 238871, Bunkyo-ku, Tokyo
  - Nippon Medical School Tama Nagayama Hospital /ID# 273428, Tama-shi, Tokyo
  - University of Yamanashi Hospital /ID# 238642, Chuo-shi, Yamanashi
  - Hayashi eye hospital /ID# 267604, Fukuoka

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=1833-201-407